CLINICAL TRIAL: NCT06081712
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Multiple Oral Doses of TNP-2198 Capsules in Asymptomatic Subjects With Helicobacter Pylori Infection
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of TNP-2198 Capsules in Asymptomatic Participants With Helicobacter Pylori Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2198-03
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Multiple Ascending Doses Cohort 1 (Experimental): TNP-2198 Capsules 200mg, BID, for 14days
  Interventions: Drug: TNP-2198; Drug: TNP-2198 Placebo
- Multiple Ascending Doses Cohort 2 (Experimental): TNP-2198 Capsules 400mg,BID, for 14days
  Interventions: Drug: TNP-2198; Drug: TNP-2198 Placebo
- Multiple Ascending Doses Cohort 3 (Experimental): TNP-2198 Capsules 600mg,BID, for 14days
  Interventions: Drug: TNP-2198; Drug: TNP-2198 Placebo

INTERVENTIONS:
Drug: TNP-2198 — TNP-2198 capsules/placebo were administered orally twice daily (BID, at 7:00 ± 1 hour in the morning and 19:00 ± 1 hour in the evening) in the fasted state for consecutive 14 days, and the last dose was taken at 7:00 am (±1 hour) on Day 15 in the fasted state, and breakfast or dinner should not be taken within 30 minutes after each dose.
  Other Names: Rifasutenizol
Drug: TNP-2198 Placebo — TNP-2198 capsules/placebo were administered orally twice daily (BID, at 7:00 ± 1 hour in the morning and 19:00 ± 1 hour in the evening) in the fasted state for consecutive 14 days, and the last dose was taken at 7:00 am (±1 hour) on Day 15 in the fasted state, and breakfast or dinner should not be taken within 30 minutes after each dose.

SUMMARY:
This study was a Phase 1, single-center, randomized, double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, and preliminary Helicobacter Pylori eradication efficacy of TNP-2198 capsules.

ELIGIBILITY:
Inclusion Criteria:

* Those signed the informed consent form and fully understood the study contents, process and possible adverse reactions before participation in the study;
* Those are able to complete the study according to the requirements in the study protocol;
* Those (including the partner) are willing to use effective contraceptions from the screening up to 6 months after the last dose of study drug;
* Male and female subjects aged 18-55 years (inclusive);
* Male subjects no less than 50 kg and female subjects no less than 45 kg. Body mass index (BMI) = body weight (kg)/height2 (m2); BMI: 18-28kg/m2 (inclusive);
* Health status: no clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system diseases, mental disorders or metabolic abnormalities;
* Normal results or clinically insignificant abnormal results in physical examinations and vital sign assessment;
* Positive result of 14C urea breath test (UBT).

Exclusion Criteria:

* Average daily consumption of more than 5 cigarettes within 3 months before the study;
* Allergic constitution (allergy to multiple drugs and food);
* History of drug and/or alcohol abuse (mean consumption of ≥ 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine);
* History of Helicobacter Pylori eradication;
* Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
* Using any drug that changes liver enzyme activity within 28 days prior to screening;
* Using any prescription drug, over-the-counter drug, any vitamin product, or herbal medicine within 14 days prior to screening;
* Taking special diet (including dragon fruit, mango, grapefruit, etc.) or strenuous exercise, or having other factors that affect drug absorption, distribution, metabolism, excretion, etc., within 2 weeks prior to screening;
* Significant changes in diet or exercise habits recently;
* Administration of any other study drug or participation in any drug clinical study within 3 months before administration of the study drug;
* With difficulty in swallowing or history of any gastrointestinal diseases that affect drug absorption;
* With any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* With clinically significant ECG abnormalities;
* Female subjects who are lactating or having positive serum pregnancy test during screening or during the study;
* With symptoms or previous history of cardiovascular, digestive, respiratory, urinary, neurological, hematologic, immunological, endocrine system diseases, tumor, or psychiatric diseases;
* Clinically significant abnormalities in clinical laboratory tests, or other clinically significant findings (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, or cardiovascular disease);
* Positive viral hepatitis (including hepatitis B and C), HIV antigen/antibody, treponema pallidum antibody;
* Acute illness or concomitant medication from the time of signing the informed consent to the time of study medication;
* Intake of chocolate, any caffeine- or xanthine-containing food or drink within 48 hours prior to administration of study drug;
* Intake of any alcohol-containing product within 48 hours before administration of study drug;
* Positive urine drug screening or history of drug abuse or drug addiction within the past 5 years;
* Other conditions that, in the opinion of the investigator, make the patient participating in this study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events(AEs) | up to 17 days
  The percentage of subjects with at least one AEs.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from the First Dose Extrapolated to Infinity (AUC0-∞) | Day 1,Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 14, Day 15
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2198 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from the First Dose to the Last Measurable Concentration (AUC 0-last) | Day 1,Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 14, Day 15
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay. Plasma PK parameters of TNP-2198 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Maximum Observed Plasma Concentration (Cmax) of TNP-2198 | Day 1,Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 14, Day 15
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: TenNor Clinical Trials, Study Director — TenNor
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Liu Y, Wang M, Gao L, Liu J, Zhang H, Wu M, Chen H, Lou J, Wang J, Chen J, Geng G, Ma Z, Ding Y. Safety, pharmacokinetics, and efficacy of rifasutenizol, a novel dual-targeted antibacterial agent in healthy participants and patients in China with Helicobacter pylori infection: four randomised clinical trials. Lancet Infect Dis. 2024 Jun;24(6):650-664. doi: 10.1016/S1473-3099(24)00003-3. Epub 2024 Feb 12. PMID 38359854